CLINICAL TRIAL: NCT01445509
Title: A Phase I Study of Dasatinib in Combination With Bevacizumab in Advanced Solid Tumors
Brief Title: Dasatinib in Combination With Bevacizumab to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 090019; 09-C-0019; NCT00792545 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01-13

CONDITIONS: Solid Tumors
Keywords: Angiogenesis; VEGF; SRC; Targeted Therapy; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Dasatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Group 1 will receive dasatinib and bevacizumab together at the start of study in a dose escalation fashion
  Interventions: Drug: Bevacizumab; Drug: Dasatinib
- Arm 2 (Experimental): Group 2 will be randomized as to which agent they receive for cycle one. Cycles 2 and beyond are treated using both agents.
  Interventions: Drug: Bevacizumab; Drug: Dasatinib

INTERVENTIONS:
Drug: Bevacizumab — Once the MTD of dasatinib with bevacizumab 5 mg/kg IV every two weeks is determined, one final dose level will be accrued with that MTD dose of dasatinib with bevacizumab at 10 mg/kg IV every two weeks in order to determine if we can safely escalate bevacizumab to full dose with dasatinib concurrently.
Drug: Dasatinib — We will start dasatinib at 50 mg PO QD which is less than half the recommended Phase 2 dose as well as bevacizumab at 5 mg/kg IV every two weeks, which is half the single agent dose. If this is well-tolerated, study drugs will be escalated per schema to maximize the dose of dasatinib when given concurrently.

SUMMARY:
Background:

* Bevacizumab inhibits blood vessel growth in cancer cells by blocking a growth factor called VEGF. Dasatinib inhibits the action of proteins called tyrosine kinases, which promote and stimulate blood vessel formation and cancer growth and spread.
* Using the two drugs in combination may provide a more effective cancer treatment than either drug used alone.
* Both drugs have been approved by the Food and Drug Administration for different cancer types, but their use in combination sis experimental.

Objectives:

- To determine the highest doses of the combination of dasatinib and bevacizumab that can be safely given to patients with different cancers and to find out what effects, good and bad, these drugs may have on the patient and the disease.

Eligibility:

- Adult patients with an advanced solid tumor cancer that cannot be treated successfully with standard therapies.

Design:

* Patients in Group 1 receive dasatinib and bevacizumab together throughout the study. The dose is increased in successive groups of three to six patients until the optimum safe dose is determined. Patients take dasatinib by mouth once a day and receive bevacizumab as an infusion through a vein once every 2 weeks in 28-day treatment cycles.
* Patients in Group 2 are randomly assigned to receive either dasatinib or bevacizumab for cycle one, and then both drugs for all subsequent cycles. The drug doses are based on the optimum doses found in Group 1 patients.
* Patients have a physical examination and blood and urine tests every 2 weeks for cycles 1 and 2, and then every 4 weeks for the duration of treatment.
* Patients have CT or MRI scans or another imaging test such as ultrasound every 8 weeks to monitor the cancer s response to treatment.
* Tumor biopsies are obtained from patients in Group 2 before treatment, 2 weeks into the first treatment cycle, and 2 weeks into the second cycle.
* Dynamic, contrast-enhanced MRI (DCE-MRI) tests are done on patients in Group 2 before treatment, 2 weeks into the first cycle and 4 weeks into the second cycle. This MRI test uses a special non-radioactive dye that shows blood flow in a certain part of the body.
* For patients who have been on the study over 2 years, the cycle may be lengthened to 6 or 8 weeks at the discretion of the investigator.

DETAILED DESCRIPTION:
BACKGROUND:

Dasatinib is an inhibitor of SRC family kinases, BCR-ABL, c-KIT, EPHA2 and PDGF beta receptor.

Bevacizumab is a humanized IgG1 monoclonal antibody (MAb) that binds all biologically active isoforms of human vascular endothelial growth factor (VEGF, or VEGF-A) with high affinity (k(d) = to 1.1nM).

This Phase I trial is open to patients with all solid tumors.

OBJECTIVES:

Determine the safety and toxicity of the combination of dasatinib and bevacizumab.

Determine biochemical changes in the src-FAK and src-PLC-gamma. and VEGF signal transduction pathways in tumor and stromal cells in response to treatment at the MTD, in a pilot fashion, if those changes are statistically significant.

ELIGIBILITY:

Adults with histologically documented solid tumor malignancy that is metastatic or unresectable and for which standard curative therapies do not exist or are no longer effective.

Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.

All patients enrolling in Group 2 must have at least one lesion amenable to biopsy.

ECOG performance status 0 or 1 and adequate organ and marrow function.

DESIGN:

Group 1 will receive dasatinib and bevacizumab together at the start of study in a dose escalation fashion.

Group 2 will be randomized as to which agent they receive for cycle one. Cycles 2 and beyond are treated using both agents.

Tumor biopsies will be obtained from patients in Group 2 before treatment, two weeks into mono-therapy, and two weeks into combinatorial therapy.

DCE-MRI studies will be obtained on patients in Group 2 before treatment, two weeks into monotherapy, four weeks into monotherapy, and two weeks into combinatorial therapy.

Patients will be evaluated for toxicity in clinic every 2 weeks for Cycles 1 and 2, and then every 4 weeks. For patients who have been on the study over 2 years, the cycle may be lengthened to 6 or 8 weeks at the discretion of the investigator.

Patients will be evaluated for response every 8 weeks using the RECIST criteria. After patients have completed 2 or more years on study, the interval may be lengthened to 12 or 16 weeks at the discretion of the investigator.

Approximately 48 patients will be needed to achieve the objectives of the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a solid tumor malignancy that is metastatic or unresectable and for which standard curative therapies do not exist or are no longer effective.

  --Patients must have histological documentation of cancer confirmed in the Laboratory of Pathology/NCI.
* Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks. Patients who were receiving mitomycin C, nitrosoureas, bevacizumab or carboplatin must be 6 weeks from the last administration of chemotherapy. Patients with prostate cancer must continue to receive LHRH agonist (unless orchiectomy has been performed). Patients should not be receiving complementary/alternative therapy while on study. Any patient who has undergone therapy with a monoclonal antibody must be at least 4 weeks from the last treatment.
* All patients enrolling in group 2 must have at least one lesion deemed safe to biopsy and be willing to undergo the three mandatory biopsies. This determination will be made by a member of the interventional radiology team or surgical associate investigator and an associate investigator. This requirement is not necessary for patients in group 1.
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of dasatinib in combination with bevacizumab in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric phase 1 combination trials.
* ECOG performance status 0 or 1. ECOG performance status of 2 will be considered on a case by case basis with a focused assessment on risk of perforation.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function as defined below:

  * Inclusion criteria laboratory values
  * Leukocytes >3,000/microl
  * Hemoglobin >= 10g/dl
  * Absolute neutrophil count >1,200/microl
  * Platelets >100,000/microl
  * total bilirubin <=1.5 X institutional upper limits of normal in the absence of Gilbert's syndrome
  * AST(SGOT) and ALT(SGPT) <=2.5 X institutional upper limit of normal
  * creatinine <=1.5 mg/dL OR Creatinine clearance >45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
  * Activated partial thromboplastin time (PTT) <= 1.25 x institutional upper limits of normal in the absence of lupus anticoagulant
  * Prothrombin Time (PT) OR INR <= 1.25 x institutional upper limits of normal
  * Spot Urine Protein Creatinine Ratio <=0.5; If result is 0.5 or more, a 24-hour urine for protein excretion must be <=1000mg
* Patients must have recovered from toxicity related to prior therapy to at least CTEP grade 1 (defined by CTCAE 4.0). Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis by the Principal Investigator.
* As the effect of dasatinib and bevacizumab in combination on the developing human fetus is not known, women of child-bearing potential and men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 3 months after completion. Pregnant women will not be eligible for study.
* Ability to understand and the willingness to sign a written informed consent document.
* Evaluable disease or measurable disease of >= 1 cm.
* Patients may not have any clinically significant cardiovascular disease including the following:

  * myocardial infarction or ventricular tachyarrhythmia within 6 months
  * prolonged QTc >=480 msec (Fridericia correction)
  * ejection fraction less than institutional normal
  * major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator. Patients with underlying cardiopulmonary dysfunction should be excluded from the

study.

EXCLUSION CRITERIA:

* Brain metastases

  * Patients who have a history of remote CNS metastases that have undergone "curative therapy" by radiation therapy, gamma knife therapy, or surgery and have remained without recurrence for a period of >=6 months will be eligible.
  * CNS imaging will not be mandated for all patients. However, if there is clinical suspicion of CNS involvement, a contrast CT or MRI of the brain will be required. Screening CNS scans should be required for certain tumor types with relatively high risk of CNS metastases, including but not limited to melanoma, renal cell carcinoma, breast, lung.
* Thrombotic or embolic events within the past 6 months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism, unstable angina, or myocardial infarction. Patients with recent (< 3 month history) of venous thrombotic events will be considered on a case by case basis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (AHA Class II or worse), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

  * Patients with evidence of active infection must have completed antibiotic therapy and be without clinical or laboratory evidence of infection for seven days after treatment has concluded.
  * QTc prolongation (defined as a QTc interval equal to or greater than 480 msecs) or other clinically significant EKG abnormalities
  * Patients may not have any clinically significant cardiovascular disease including the following:
  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged QTc >= 480msec (Fridericia correction)
  * Ejection fraction less than institutional normal (should be done if clinically indicated and for patients with congestive heart failure on medication)
  * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients who have an active pleural effusion may be considered if tapped prior to study. Patients with pleural effusions that are too small to be removed may be considered on a case by case basis. Patients with a Grade 2, asymptomatic pericardial effusion found incidentally on imaging studies may be considered on a case by case basis.
  * Dasatinib is metabolized primarily by the CYP3A4 liver enzyme. Consideration should be given to using alternative medications not impacting CYP3A4 while on dasatinib therapy.
  * Patients may not be receiving any prohibited potent CYP3A4 inhibitors. For these drugs, a wash-out period of >= 7 days is required prior to starting dasatinib treatment.
  * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes. A wash-out period of >= 7 days is required for the following drugs prior to starting dasatinib treatment:

    * Quinidine, procainamide, disopyramide
    * Amiodarone, sotalol, ibutilide, dofetilide
    * Erythromycin, clarithromycin
    * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
    * Cisapride, bepridil, droperidol, methadone, arsenic, chlorquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with dasatinib, bevacizumab, and/or the combination. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who have been treated with dasatinib (or any other Src-family kinase inhibitors) will be excluded
* Hypertension defined as systolic blood pressure >140 mmHg or diastolic pressure >= 90 mmHg despite optimal medical management.
* Proteinuria defined as a spot urine analysis for protein creatinine ratio (UPC) of > 1.0
* Therapeutic anticoagulation with coumadin, heparins, or heparinoids. Prophylaxis doses are permitted.
* Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months of fracture. History of abdominal fistula, major surgery, bowel obstruction, or intra-abdominal abscesses within 28 days will be excluded. Any patient with history of gastrointestinal perforation will be excluded due to possibility of increased risk of perforation with bevacizumab.
* Evidence of bleeding diathesis
* Impairment of swallowing that would preclude administration of dasatinib.
* History of hemoptysis or surgery within the past 28 days.
* Patients with squamous cell carcinoma of the lungs will be excluded due to risk of fatal pulmonary hemorrhage. If a patient has a history of any type primary lung cancer and hemoptysis, they will be excluded.
* History of high grade varices.
* Use of herbal supplements are not permitted within 7 days of trial commencement and on study. Vitamin supplement (above a typical single multi-vitamin) usage is discouraged unless clearly indicated by an existing medical condition. An Associate or Principal Investigator will have the discretion regarding which vitamin supplements are permitted.
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies.
* Use of any other concurrent investigational agents for treatment or anticancer agents including hormonal therapy, except in the case of prostate cancer patients who are being treated with LHRH agonist at the time of trial entry
* Pregnant women are excluded from this study because bevacizumab is an antibody to VEGF with the potential for teratogenic or abortifacient effects. Dasatinib is a potential teratogen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother bevacizumab or dasatinib, breastfeeding should be discontinued if the mother is treated on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-12-29 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Determine the toxicity profile of the combination of dasatinib and bevacizumab | end of treatment
  A safety and toxicity profile of the combination of dasatinib and bevacizumab
Maximjum Tolerated Dose (MTD) of the combination of dasatinib and bevacizumab | every 2 weeks for cycles 1 and 2; then every 4 weeks
  Determine the MTD of the combination of dasatinib and bevacizumab
Estimates of biochemical changes in the src-FAK and src-PLC- and VEGF signal transduction pathways | at the MTD
  A describe of biochemical changes in the src-FAK and src-PLC- and VEGF signal transduction pathways in tumor and stromal cells in response to treatment for Group 2.

SECONDARY OUTCOMES:
Efficacy of the combination of bevacizumab and dasatinib. | End of treatment
  Determine preliminary evidence of efficacy of the combination of bevacizumab and dasatinib. Determine biochemical changes in the src-FAC and src-PLC-y and VEGF signal transduction pathways in tumor and stromal cells in response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Lipkowitz, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avizienyte E, Wyke AW, Jones RJ, McLean GW, Westhoff MA, Brunton VG, Frame MC. Src-induced de-regulation of E-cadherin in colon cancer cells requires integrin signalling. Nat Cell Biol. 2002 Aug;4(8):632-8. doi: 10.1038/ncb829. PMID 12134161
- [Background] Burger RA, Sill MW, Monk BJ, Greer BE, Sorosky JI. Phase II trial of bevacizumab in persistent or recurrent epithelial ovarian cancer or primary peritoneal cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Nov 20;25(33):5165-71. doi: 10.1200/JCO.2007.11.5345. PMID 18024863
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0019.html